CLINICAL TRIAL: NCT05724420
Title: Evaluation of a Formal Resilience Curriculum for Novice Physicians-in-training on Self-reported Resilience: a Randomized Controlled Trial
Brief Title: STRIVE - Resilience Curriculum for Novice Physicians-In-Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Sonja Payne, Assistant Professor, Consultant Anesthesiologist, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 13156
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Stress, Emotional
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial with a 1:1 allocation ratio between intervention (STRIVE course) and control groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Sequence generation: computer-generated randomization in REDCAP program to two groups for each resident year cohort; STRIVE program and control group.
  Blinding: Post-interventional analysis will be performed by a dedicated team member blinded to the intervention assignment who will not participate in course delivery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STRIVE Group (Experimental): STRIVE is comprised of a 4-hour formal education session where participants are provided knowledge, skills, and resources specific to self-assessment for mental wellness and effective mindfulness strategies.
  High-fidelity simulation sessions are utilised to reinforce and apply mindfulness techniques learned in the formal session. Clinical scenarios are designed to be challenging and stressful.
  Interventions: Behavioral: STRIVE course delivery
- Control (No Intervention): Residents randomized to the control group will receive information regarding resilience development as per the usual standard of communication. All new residents will receive contact details of physician wellness services available at Schulich School of Medicine & Dentistry.

INTERVENTIONS:
Behavioral: STRIVE course delivery — STRIVE is adapted from the Road to Mental Readiness curriculum, developed by the Department of National Defence in Canada. It is comprised of a 4-hour formal education session where participants are provided knowledge, skills and resources specific to self-assessment for mental wellness and effective mindfulness strategies. High fidelity simulation sessions are then utilized to reinforce and apply mindfulness techniques learned in the formal session..
  Arms: STRIVE Group

SUMMARY:
The goal of this trial is to compare self-reported resilience scores in junior physicians-in-training after completion of formal resilience training. The main questions this trial aims to answer are:

* Does formal resilience training improve self-reported resilience scores?
* Does the timing of resilience training (i.e., first vs second year of residency training) impact the effect of training? All participants will be provided with resources on resilience and learner support as per usual institutional practice. The intervention group will also participate in a formal resilience training program.

Researchers will compare self-reported resilience scores 3 months after training to determine the effect of the training program.

DETAILED DESCRIPTION:
Physician wellness has gained much attention over recent years due to growing concerns regarding mental illness and burnout. The COVID-19 pandemic further highlighted the importance of physician health.

Resilience, defined as the capacity of an individual to adapt well and even thrive in the setting of adversity and stress, has been identified as an indicator of physician wellness. Resilience is a multidimensional concept that integrates personal factors, such as personality, with previous challenging experiences, leading to positive adaptation.

Simulation Training for Resilience in Various Environments (STRIVE) is an adaptation of a formal resilience curriculum developed by the Department of National Defense in Canada for military personnel. Fundamental skills learned during the course are applied and reinforced through experiential learning with high-fidelity simulation accompanied by effective debriefing.

Physicians-in-training have been identified as a population cohort with a high prevalence of burnout, depersonalization, and fatigue. Research demonstrates that institutional culture on wellbeing has a greater impact on resident satisfaction compared to the area of specialization. Therefore, we propose that institutional curricula and training in physician wellness may improve self-reported resilience in physicians-in-training.

The study will be conducted at London Health Sciences Centre, University Hospital in London, Ontario. A total of 60 participants will be recruited from the PGY-1 and PGY-2 residents from the Anesthesia and Emergency Medicine residency programs at the commencement of the academic year 2023.

The study aims to compare self-reported resilience of participants before and after the training, to determine if there is a statistically significant improvement in resilience scores, based on the CD-RISC-10 scores at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* All first- and second-year medical residents enrolled in the Schulich School of Medicine & Dentistry Anesthesia and Emergency Medicine postgraduate residency programs will be eligible to participate, regardless of age, gender, health status, or race. The respective residency program directors have approved study content and procedure.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate of the effect of formal resilience training using the STRIVE course on self-reported resilience at 3 months. | 3 months
  Self-reported resilience will be quantified using the abbreviated Connor-Davidson Resilience Scale (CD RISC-10). Scores range from 0 to 40 with a higher score indicating higher resilience.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No